CLINICAL TRIAL: NCT02791633
Title: Recovery After Emergency Laparotomy: a Prospective Observational Feasibility Study
Acronym: REmLap
Status: Completed | Type: Observational
Sponsor: Dudley Group NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: REmLap
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Quality of Life; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Quality of recovery and quality of recovery follow up questionnaires
  Other Names: WHODAS, SF36, QOR15, POMS

SUMMARY:
Observational feasibility study using Patient Reported Outcomes (PRO) to assess quality of life and 'return to normal life' up to 1 year following emergency laparotomy

DETAILED DESCRIPTION:
Regaining baseline Health Related Quality of Life (HRQoL) and returning to 'normal life' after surgery are of vital importance for patients. Knowledge of the trajectory and degree of long-term functional recovery following emergency laparotomy, including the regaining of optimal HRQoL is limited as most research relating to this field has been done in patients undergoing planned surgery. Furthermore, a comprehensive understanding of the pattern of recovery and restoration of baseline HRQoL is also important to researchers wishing to assess the full impact of interventions in order to improve outcomes following emergency laparotomy. Assessing HRQoL in this surgical population remains a challenge in the absence of a validated instrument. The investigators plan to undertake a feasibility study to assess utilisation of four patient questionnaires, well established within other surgical populations, to describe the quality of early and long-term recovery following emergency laparotomy. The investigators will utilise the QoR-15 to describe short-term (in - hospital) recovery metrics and versions of the WHO-DAS and the WHOQOL-BREF to describe longer term disability free survival and return towards baseline HRQoL. The Post-Operative Morbidity Survey (POMS) will help capture the onset of complications at different points during recovery. The study also aims to test the feasibility of assessing the impact of pre-operative co-morbidities, age, quality of peri-operative and intra-operative care, surgical indication and findings as well as post-operative complications on long-term HRQoL.

ELIGIBILITY:
Inclusion Criteria:

- >=18 years NELA Inclusion Criteria

Exclusion Criteria:

- Not willing to participate NELA Exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting NELA inclusion criteria (National Emergency Laparotomy Audit), undergoing Emergency Laparotomy at Russells Hall Hospital agreeing to participate
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Disability free survival | 1 year
  Disability free survival

SECONDARY OUTCOMES:
Change in Quality of life | 1 year
  Use of WHODAS-12, WHOQOL-BREF with specific symptom questionnaires
Impact of surgical pathology type on disability free survival | 1 year
  Impact of surgical pathology type on disability free survival
Impact of pre-operative Charlson Score on disability free survival | 1 year
  Impact of pre-operative Charlson Score on disability free survival

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Jennings, Study Director — Dudley Group NHSFT; Rajan Patel, Study Director — DGNHSFT; Faisal Baig, Study Director — DGNHSFT; Peter Waterland, Study Director — DGNHSFT
Locations (1):
- Russells Hall Hospital, Dudley, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No